CLINICAL TRIAL: NCT05915624
Title: The Effect of Pre-Surgery Tele Nursing Counseling on Anxiety and Patient Satisfaction in Same Day Surgery
Brief Title: Tele Nursing Counseling on Anxiety and Patient Satisfaction in Same Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Assoc.Prof.Ezgi Seyhan Ak (Unknown)
Responsible Party: Principal Investigator, Nasır Mehmet Özbek, Master Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IUCESEYHANAK001
Record Dates: First submitted 2023-06-10; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Ambulatory Surgical Procedures
Keywords: ambulatory surgery; anxiety; patient satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The patients in the experimental group will be given a Preoperative Patient Information Brochure prepared by the researcher when they come to the hospital for the surgery date after the voluntary informed consent form is signed. Data were collected using the Introductory Information Form and the Surgery-Specific Anxiety Scale, and counseling was provided by tele-nursing information about the surgery process one day before the surgery. Patient's Perception of Nursing Care Scale was applied before leaving the hospital after day surgery.The patients in the control group were given a Preoperative Patient Information Brochure, which was prepared by the researcher on the day of the surgery, when they came to the hospital for the surgery date after signing the voluntary informed consent form. Data were collected using the Introductory Information Form and the Surgery-Specific Anxiety Scale. Patient's Perception of Nursing Care Scale was applied before leaving the hospital after day surgery.
Who Masked: Participant
Masking Description: The participant does not know which group he/she is in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone counseling group (Experimental): After signing the voluntary informed consent form, the patients in the experimental group were given a Preoperative Patient Information Brochure, prepared by the researcher when they came to the hospital for the surgery date. Data will be collected using the Introductory Information Form and the Surgery-Specific Anxiety Scale, and counseling was provided by tele-nursing information about the surgery process one day before the surgery.
  Interventions: Other: telephone counseiling
- Control group (No Intervention): The patients in the control group were given a Preoperative Patient Information Brochure, which was prepared by the researcher on the day of the surgery, when they came to the hospital for the surgery date after signing the voluntary informed consent form.

INTERVENTIONS:
Other: telephone counseiling — One day before the operation, information was given about the operation process via tele-nursing and counseling was provided.
  Arms: telephone counseling group

SUMMARY:
The study was planned to be conducted as a randomized controlled experimental study to examine the effect of preoperative tele-nursing counseling on anxiety and patient satisfaction in same day surgery.

The main Research Hypotheses are; Preoperative tele-nursing counseling has no effect on anxiety in same day surgery.

Preoperative tele-nursing counseling has an effect on anxiety in same day surgery.

Preoperative tele-nursing counseling has no effect on patient satisfaction in same day surgery.

Preoperative tele-nursing counseling has an effect on patient satisfaction in same day surgery.

DETAILED DESCRIPTION:
Power analysis was performed using the G*Power (v3.1.7) program to determine the number of samples. The power of the study (α) was accepted as 0.05 (95% confidence level), Type 2 error probability (β) was accepted as 0.20 (80% power level) and the effect size of 0.46 in the relevant literature (Pehlivan, 2021) was taken into account, and the minimum required minimum in the groups was taken into account. It was found that taking the sample size as 74 would be sufficient. In the study, it was aimed to have a total of 148 participants, 74 for the control group and 74 for the experimental group. Considering the possible loss, the study was completed with a total of 160 patients, 80 of which were in the control group and 80 in the experimental group.

While evaluating the findings obtained in the study, SPSS (Statistical Package for the Social Sciences) version 25.0 (IBM Corp., Armonk, NY, USA) program will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old,
* Agreeing to participate in the research,
* Persons who will undergo day surgery in the field of general surgery, urology, orthopedic surgery, plastic surgery, neurosurgery,
* GKS score of 15,
* Not addicted to alcohol
* No psychiatric problems,
* Not using antipsychotic, antidepressant and anxiolytic drugs
* According to the ASA (American Society of Anesthesiologists) classification, ASA 1-2-3 -classification
* Speech and hearing impaired
* It is planned to include patients who have an open phone in the study.

Exclusion Criteria:

* Preoperative hospitalization
* Patients undergoing emergency surgery
* Patients who want to leave the study at any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Surgery-Specific Anxiety Scale | two hours before going to surgery
  It is a 5-point Likert-type scale. (1-Strongly disagree, 2-Disagree, 3-Undecided, 4-Agree, 5-Completely agree). The maximum score to be taken from the scale is 50. In the scale scoring system, the emotions experienced by the patients were collected in 3 different dimensions.
Patient's Perception of Nursing Care Scale | two hours before discharge
  It was used to measure the satisfaction level of patients with nursing care. It is required to mark one of the 15 statements that make up the scale: Agree-5, Agree a little-4, Undecided-3, Disagree-2, Strongly Disagree-1 and No response-0. The score given for each item is taken as a basis. Thus, a minimum of 15 and a maximum of 75 points can be obtained from the scale. The cut-off point of the scale is 45. Scores above the cut-off point indicate a positive attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Ezgi Seyhan Ak, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No